CLINICAL TRIAL: NCT05271331
Title: ESP Block Versus Wound Infiltration for Laminectomy: a Randomized Controlled Trial
Brief Title: ESP Block Versus Wound Infiltration for Laminectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Geraldini, Principal Investigator, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5211/AO/21
Record Dates: First submitted 2022-02-23; First posted 2022-03-09 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Opioid Use; Anesthesia, Local; Surgery
Keywords: ESP block; Laminectomy; Wound infiltration
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both arms will receive the same treatment (Wound infiltration and ESP block) after general anesthesia induction (Participant masked to intervention) Drugs will be prepared after randomization by a physician not involved in the care of the patients and not involved in the study, and labelled as WOUND INFILTRATION and ESP block. One syringe will contain local anesthetic, the other normal saline (Care Provider masked to intervention, Investigator masked to intervention) Outcome assessor will be not involved in other part of the study and will be not aware of the intervention (Outcome assessor masked to intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESP block (Experimental): Patient will receive ESP block one level above surgery with ropivacaine 0.35% 20 ml per side Patient will receive preoperative wound infiltration with Saline 40 ml
  Interventions: Drug: Wound infiltration with saline; Drug: ESP block with local anesthetic
- Wound infiltration (Active Comparator): Patient will receive ESP block one level above surgery with Saline 20 ml per side Patient will receive preoperative wound infiltration with ropivacaine 0.35% 40 ml
  Interventions: Drug: ESP block with saline; Drug: Wound infiltration with local anesthetic

INTERVENTIONS:
Drug: ESP block with saline — Bilateral ultrasound guided injection of saline in the erector spinae plane (below erector spinae plane muscle group and above the transverse process of the vertebra)
  Other Names: Erector spinae plane block
  Arms: Wound infiltration
Drug: Wound infiltration with saline — Blinded injection of saline in the skin, subcutaneous tissue and muscles at the site of surgical incision
  Arms: ESP block
Drug: ESP block with local anesthetic — Bilateral ultrasound guided injection of local anesthetic (ropivacaine 0.35%, 40ml) in the erector spinae plane (below erector spinae plane muscle group and above the tranverse process of the vertebra)
  Other Names: Erector spinae plane block
  Arms: ESP block
Drug: Wound infiltration with local anesthetic — Blinded injection of local anestetic (ropivacaine 0.35%, 40ml) in the skin, subcutaneous tissue and muscles at the site of surgical incision.
  Arms: Wound infiltration

SUMMARY:
Spinal surgery is often burdened by perioperative pain and its treatment presently represents a challenge for anesthetists. An inadequate intra and postoperative analgesic therapy leads to a delay in the mobilization of the patients, prolonged hospital stay and thromboembolic complications, as well as the onset of chronic pain syndromes . Effective pain treatment can help improve surgical outcome for patients undergoing spinal surgery. From the pathophysiological point of view pain in vertebral surgery can originate from different anatomical structures: vertebrae, discs, ligaments, dura mater, facet joints, muscles and skin-subcutis. The terminal innervation of these tissues originate from the dorsal branches of the spinal nerves, and this represents a target a multimodal approach to perioperative analgesia in vertebral surgery. Systemically administered drugs such as NSAIDs, opioids, ketamine, intravenous lidocaine could benefit from the addition of locoregional therapies such as neuraxial blocks (anesthesia peridural or subarachnoid) or as shown more recently by other anesthesia techniques locoregional ultrasound-guided In recent years the anesthesiological interest has focused on the Erector Spinae Plane Block (ESPB). First described by Forero et al, it is a paraspinal interfascial block targeting the dorsal and ventral branches of the spinal nerves just after their emergence from the spinal cord. In the ultrasound-guided technique the local anesthetic is injected between the deep fascia of the muscle itself and the transverse processes of the vertebrae at the level interested. The aim of this study is to evaluate the efficacy of ESPB when compared to wound infiltration in patients undergoing laminectomy

ELIGIBILITY:
Inclusion Criteria:

-Planned 1 or 2 level surgical laminectomy

Exclusion Criteria:

* Allergy to local anesthetics
* Refusal of consent
* Uncompensated cardiopathies, nephropathies, liver disease or peripheral neuropathies
* Hemopathies that predispose to bleeding
* Gastrointestinal ulcer or bleeding
* Local infection
* Psychiatric or neurological disorders (except those attributed to primary disease for which intervention is planned) History of abuse (or use in the 24 hours prior to surgery) Alcohol addiction ASA > 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Tramadol consumption | Evaluated from extubation for the first post-operative 24 hours
  Postoperative tramadol consumption

SECONDARY OUTCOMES:
Pain 0 hours | At extubation
  Pain measured with Numeric Rating Scale (0-10)
Pain 6 hours | 6 hours after end of surgery
  Pain measured with Numeric Rating Scale (0-10)
Pain 12 hours | 12 hours after end of surgery
  Pain measured with Numeric Rating Scale (0-10)
Pain 24 hours | 24 hours after end of surgery
  Pain measured with Numeric Rating Scale (0-10)
Time to first analgesic requirement | 24 hours after end of surgery
  Time in minutes to first analgesic requirement
Incidence of post operative nausea-vomiting | 24 hours after end of surgery
  Incidence of post operative nausea-vomiting
Incidence of post operative respiratory depression | 24 hours after end of surgery
  Incidence of post operative respiratory depression
Incidence of post operative pruritus | 24 hours after end of surgery
  Incidence of post operative pruritus
Incidence of post operative motor block | 24 hours after end of surgery
  Incidence of post operative motor block
Intraoperative opioid consumption | At extubation
  Intraoperative difference in consumption of fentanyl.
Evaluation of patient satisfaction | 24 hours after end of surgery
  Evaluation of patient satisfaction of analgesia on a numeric rating score from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Geraldini, MD, Principal Investigator — University Hospital of Padova
Locations (1):
- University Hospital of Padova, Padua, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared on reasonable request after ethical committee request examination